CLINICAL TRIAL: NCT05718882
Title: Safety and Efficacy of Lenvatinib Combined With VIC-1911 in the Treatment of Lenvatinib-unresponsive or Lenvatinib-resistant Hepatocellular Carcinoma
Brief Title: Lenvatinib Plus VIC-1911 in Lenvatinib-unresponsive or Lenvatinib-resistant HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renji-LY2022-024-b
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Resistant Cancer
Keywords: Aurora A kinase inhibitor
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Bayesian Optimal Interval design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib plus VIC-1911 combination therapy (Experimental): Subjects with lenvatinib unresponsive or lenvatinib resistant hepatocellular HCC will receive Lenvatinib plus VIC-1911 combination therapy.
  Interventions: Drug: Lenvatinib Oral Product Plus VIC1911

INTERVENTIONS:
Drug: Lenvatinib Oral Product Plus VIC1911 — Lenvatinib: 8mg/day (≤ 60Kg), oral. VIC-1911:Groups were divided: 100mg bid（DL1, dose level 1）; 150mg bid（DL2）; 200mg bid(DL3), oral. 50mg bid is defined as DL(-1), 250mg bid is defined as DL(+1). A Bayesian Optimal Interval design schema will be followed to establish the maximum tolerated dose (MTD) of lenvatinib plus VIC-1911 combination and RP2D of VIC-1911 in HCC patients. The study would follow the Bayesian Optimal Interval Design with level size of 2 patients. The R package "BOIN" is available from CRAN.
  Other Names: aurora kinase A inhibitor

SUMMARY:
This is a prospective clinical study aiming to test the safety and efficacy of lenvatinib in combination with Aurora kinase A inhibitor VIC-1911 in participate with lenvatinib-unresponsive or lenvatinib-resistant hepatocellular carcinoma(HCC).

ELIGIBILITY:
Inclusion Criteria:

(1) Unlimited gender, aged 18-75 years; (2) Meets American Association for the Study of Liver Diseases (AASLD) or European Association for the Study of the Liver (EASL) clinical diagnostic criteria of hepatocellular carcinoma; (3) Barcelona Clinic Liver Cancer (BCLC) Stage C, and there is at least one measurable tumor in the liver (long diameter ≥ 1cm);(4) Lenvatinib unresponsive or lenvatinib resistant after standard treatment; (5) Child-Pugh A or scored 7 B; (6) Eastern Cooperative Oncology Group performance status score <= 1; (7) Platelet count >= 60x10^9/L, Prothrombin time prolonged <= 6 seconds.

Exclusion Criteria:

(1) Uncorrectable coagulopathy with obvious bleeding tendency; (2) Patients need long-term anticoagulant or anti platelet therapy and cannot stop the drugs; (3) Patients with unstable or active ulcer or gastrointestinal bleeding; (4) Heart disease requiring treatment or not well controlled high blood pressure; (5) Hepatic encephalopathy or refractory ascites requiring treatment; (6) There is a clear active infection; (7) Receiving radiotherapy/chemotherapy/interventional therapy for tumor within 4 weeks before the start of the study; (8) Severe insufficiency of important organs, such as severe cardiopulmonary insufficiency; (9) Other accompanying anti-tumor treatments; (10) The investigator assessed that the patient was unable or unwilling to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months after the last subject is enrolled.
  Length of time from the start of combination therapy to progression of disease or death

SECONDARY OUTCOMES:
Overall survival | 6 months after the last subject is enrolled
  Length of time from the date of first dose of combination therapy to date of death from any cause or latest follow-up
Safety endpoint | 6 months after the last subject is enrolled
  Statistically describe the proportion of adverse events after treatment for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Qiang XIA, Study Chair — Dept. Liver Surgery, Renji Hospital, School of Medicine, SJTU
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China